CLINICAL TRIAL: NCT02267681
Title: The Effects of Fentanyl and Alfentanil as an Adjunct to Propofol on Cognitive Functions for Sedation in Colonoscopy
Brief Title: Opioid Effects on Cognitive Function Following Colonoscopy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Perihan Ekmekçi (Other)
Responsible Party: Sponsor-Investigator, Perihan Ekmekçi, Assistant Professor, Ufuk University
Organization: Ufuk University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: Ufuk University
Record Dates: First submitted 2014-10-14; First posted 2014-10-17 (Estimated); Last update posted 2016-06-29 (Estimated); Status verified 2016-06

CONDITIONS: Digestive System Diseases; Disorientation
MeSH Terms: conditions — Digestive System Diseases; Confusion | interventions — Fentanyl; Alfentanil; Propofol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group A (Experimental): The patients in Group A will be given 100 mcg/kg/min propofol infusion and 10 mcg/kg loading dose of alfentanil and 5 mcg/kg additional bolus of alfentanil whenever FPS (Faces Pain Scale) is greater than 3 or the patients can not tolerate the procedure.
  Interventions: Drug: Alfentanil; Drug: Propofol
- Group F (Experimental): The patients in Group F will be given 100 mcg/kg/min propofol infusion and 1 mcg/kg loading dose of fentanyl and 5 mcg/kg additional bolus of fentanyl whenever FPS (Faces Pain Scale) is greater than 3 or the patients can not tolerate the procedure.
  Interventions: Drug: Fentanyl; Drug: Propofol
- Group P (Active Comparator): Group P is designated as the control group and the patients will be given 100mcg/kg/min infusion and sedation will be achieved via 1 mg/kg propofol loading dose and 0.5 mg/kg propofol additional bolus will be given whenever the patients can not tolerate the procedure or FPS is greater than 3.
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Fentanyl — Intravenous fentanyl for sedation/analgesia
  Other Names: Talinat
  Arms: Group F
Drug: Alfentanil — Intravenous alfentanyl for sedation/analgesia
  Other Names: Rapifen
  Arms: Group A
Drug: Propofol — Intravenous propofol for sedation
  Other Names: Diprivan

SUMMARY:
This study aims to compare the effects of fentanyl and alfentanil on postprocedural cognitive function in elective endoscopy.

150 patients will be enrolled in the study. Patients meeting eligibility criteria will be randomly allocated to three groups.

The patients in Group A will be given propofol and alfentanil. The patients in Group F will be given propofol and fentanyl. Group P is designated as the control group and the patients will be given propofol for sedation.

Awareness, vital signs and pain will be evaluated. Side effects will be recorded. Patient and endoscopist satisfaction will be evaluated.

DETAILED DESCRIPTION:
In this study we aimed to compare the effects of sedation provided by propofol with the addition of the short-acting opioid alfentanil and long-acting opioid fentanyl on cognitive functions, pain, side effects during the procedure and the endoscopist and patient satisfaction.

Following the approval of Kırıkkale University ethics committee, 150 patients ages between 18 and 65 ASA I-III scheduled for elective endoscopy and colonoscopy will be enrolled in the study.

After obtaining written informed consent, APAIS (The Amsterdam Preoperative Anxiety and Information Scale) and MMTS (Mini Mental Test Scoring) tests will given to patients. Following TDT (Trieger Dot Test) and DSST (Digit Symbol Substitution Test), the patients will be randomly allocated to either Propofol-Alfentanil (Group A), Propofol-Fentanyl (Group F) or Propofol-Control (Group P) which consists of 50 patients each.

The patients in Group A will be given 100 mcg/kg/min propofol infusion and 10 mcg/kg loading dose of alfentanil and 5 mcg/kg additional bolus of alfentanil whenever FPS (Faces Pain Scale) is greater than 3 or the patients can not tolerate the procedure.

The patients in Group F will be given 100 mcg/kg/min propofol infusion and 1 mcg/kg loading dose of fentanyl and 5 mcg/kg additional bolus of fentanyl whenever FPS (Faces Pain Scale) is greater than 3 or the patients could not tolerate the procedure.

Group P is designated as the control group and the patients will be given 100mcg/kg/min infusion and sedation will be achieved via 1 mg/kg propofol loading dose and 0.5 mg/kg propofol additional bolus will be given whenever the patients can not tolerate the procedure or FPS is greater than 3.

BIS values, mean arterial pressures, heart rates, peripheral oxygen saturations will be recorded in all three groups. FPS and VAS (Visual Analogue Scale) values will be evaluated.

Patients with intraprocedural desaturation, hypo- or hypertension, brady- or tachycardia, nausea, vomiting and apnea will be recorded. Total amounts of drugs administered will be recorded.

Infusions will be ceased at the end of the procedure and the time for OAAS/S to exceed 3 will be recorded and TDT and DSST will be repeated at 5, 15 and 30th minutes. Patient and endoscopist satisfaction will be evaluated in all cases.

ELIGIBILITY:
Inclusion Criteria:

* Ages between 18-65
* American Society of Anesthesiologists classification I-III
* Patients scheduled to undergo elective colonoscopy or endoscopy and colonoscopy

Exclusion Criteria:

* Patients younger than 18 or older than 65
* Mini mental test score < 26
* APAIS (The Amsterdam Preoperative Anxiety and Information Scale) >10
* Serious systemic disease
* Neuropsychiatric disorder
* Chronic alcohol abuse
* Morbid obesity
* History of anesthesia in the last 7 days
* Known allergy to study drugs

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2014-10; Primary Completion 2016-05 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
cognitive dysfunction | during the 30 minutes after the termination of the procedure
  as evaluated using Trieger dot test,Mini mental test and Digit symbol substitution test

SECONDARY OUTCOMES:
Patient and endoscopist satisfaction | following the procedure
  as evaluated using a 5-point Likert scale
Pain | during the 30 minutes after the termination of the procedure
  as evaluated using VAS score
Side effects | during the 30 minutes after the termination of the procedure
  hypotension, hypertension, bradycardia, tachycardia, apnea, nausea and vomiting

CONTACTS AND LOCATIONS:
Overall Officials: Perihan Ekmekçi, MD, Principal Investigator — Ufuk University
Locations (1):
- Ufuk University Dr Rıdvan Ege Hospital, Ankara, Turkey (Türkiye)

REFERENCES:
- [Background] Froehlich F, Gonvers JJ, Fried M. Conscious sedation, clinically relevant complications and monitoring of endoscopy: results of a nationwide survey in Switzerland. Endoscopy. 1994 Feb;26(2):231-4. doi: 10.1055/s-2007-1008949. PMID 8026371
- [Background] Turk HS, Aydogmus M, Unsal O, Koksal HM, Acik ME, Oba S. Sedation-analgesia in elective colonoscopy: propofol-fentanyl versus propofol-alfentanil. Braz J Anesthesiol. 2013 Jul-Aug;63(4):352-7. doi: 10.1016/j.bjane.2012.07.007. Epub 2013 Aug 13. PMID 24565243